CLINICAL TRIAL: NCT01804556
Title: The Effects of the Myofascial Trigger Point Injections on Pain and Sleep Disturbance in Patients With Nocturnal Leg Cramps With Trigger Points on Gastrocnemius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0197
Record Dates: First submitted 2013-03-03; First posted 2013-03-05 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Nocturnal Leg Cramps
Keywords: muscle cramps, trigger points, sleep disturbance
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Muscle Cramp; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myofascial trigger point injection (Other): Myofascial trigger point injection on gastrocnemius muscle
  Interventions: Procedure: Myofascial trigger point injections on gastrocnemius muscle

INTERVENTIONS:
Procedure: Myofascial trigger point injections on gastrocnemius muscle — On the first visit (T0), we record numeric rating scale (NRS), the frequency of cramps and insomnia severity index using questionnaires. Then we check trigger points of gastrocnemius muscle and inject lidocaine 1 ~ 2 ml each up to four points. One week later (T1) we record numeric rating scale (NRS), the frequency of cramps and insomnia severity index again, check trigger points, and if any, inject lidocaine. If the patient do not come, we get numeric rating scale (NRS), the frequency of cramps and insomnia severity index over the telephone. Two weeks after the first visit (T2), we repeat the procedure of the first visit (T0). And four weeks after the first visit (T3) we record numeric rating scale (NRS), the frequency of cramps and insomnia severity index through face-to-face interview or by telephone.

SUMMARY:
Nocturnal leg cramps is involuntary strong contraction of leg muscle, mostly in calves. It occurs suddenly and induces pain. Patients with frequent nocturnal leg cramps suffer from sleep disturbance in company with pain. In the present study, we examined the effects of the myofascial trigger point injections, which are known to be helpful for ease of nocturnal leg cramps, on pain and sleep disturbance in patients with nocturnal leg cramps with trigger points on gastrocnemius muscle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-80 years of age) scheduled for myofascial trigger point injections on gastrocnemius muscle due to nocturnal leg cramps at least once a week

Exclusion Criteria:

* Patients with no trigger points on gastrocnemius muscle,
* electrolyte abnormality,
* congenital musculoskeletal disorder,
* local or systemic infection, bleeding disorder or the use of anticoagulation medications,
* known allergy of local anesthetics, or the use of hypnotics or sedatives in the last 1 month

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain score | 4 weeks
  Pain score measured by numeric rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025